CLINICAL TRIAL: NCT02272231
Title: Pathogenesis of Bacterial Vaginosis in Women Who Have Sex With Women
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University of Mississippi Medical Center (Other); Louisiana State University Health Sciences Center in New Orleans (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Dr. Christina Muzny, Associate Professor - Med-Infectious Disease, University of Alabama at Birmingham
Other Study IDs: F131127001
Record Dates: First submitted 2014-10-20; First posted 2014-10-22 (Estimated); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Vaginosis, Bacterial
Keywords: women's health; vaginosis, bacterial; african americans
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Self-collected vaginal swabs from women participating in this study will be stored for future research purposes related to the study of the vaginal microbiome.
Oversight: Data Monitoring Committee: No

SUMMARY:
The objectives of this study are to: (1) use cultivation-independent molecular methods to determine the sequence of microbiological events culminating in bacterial vaginosis (BV) among sexually active African American women who have sex with women (AAWSW) and (2) determine if specific Gardnerella vaginalis oligotypes are associated with the development of BV among sexually active AAWSW.

DETAILED DESCRIPTION:
Bacterial vaginosis (BV) is the most common cause of vaginal discharge in the U.S. It is associated with adverse outcomes including preterm birth, pelvic inflammatory disease, and increased risk of acquisition and transmission of sexually transmitted infections (STIs), including HIV. Microbiologically, BV is characterized by depletion of lactobacilli that comprise the normal vaginal flora and increases in facultative (Gardnerella vaginalis; GV) and strict anaerobes.

Three out of four Amsel criteria are necessary for the clinical diagnosis of BV and include (1) homogeneous, thin, grayish-white vaginal discharge, (2) vaginal pH >4.5, (3) positive whiff-amine test, and (4) clue cells present on a wet mount of vaginal fluid. BV diagnosis, however, is based most rigorously on Nugent scoring of a Gram stain of vaginal secretions. Optimal vaginal flora, indicative of a predominance of lactobacilli, is represented by a Nugent score of 0-3. Abnormal vaginal flora includes not only what is currently defined as BV (Nugent score 7-10) but also what is referred to as intermediate flora (Nugent score 4-6). For reasons not well understood, BV is very common among women who have sex with women (WSW), perhaps more so than among heterosexual women. Risks for prevalent BV among WSW have included higher numbers of lifetime female sexual partners, shared use of vaginally inserted sex toys, and oral-anal sex. In addition, WSW in monogamous sexual partnerships have a high concordance for the presence or absence of BV. These data support the hypothesis that BV is sexually transmitted.

It is well accepted that BV is caused by a synergistic relationship between a large number of microorganisms including GV and other anaerobics (i.e. BV-associated bacteria; BVAB) however the trigger which initiates these alterations is debated. It is unknown whether BV results from acquisition of GV as the "founder" organism which subsequently leads to the complex changes in the vaginal microbiota associated with BV or whether BV is transmitted as a polymicrobial consortium. GV, as a facultative anaerobe, may be better able to tolerate the high oxidation-reduction (redox) potential of the healthy vaginal microbiome, unlike strict anaerobes. Similar to facultative anaerobes involved in the initiation of oral disease, it is possible that GV, through its metabolic pathways and ability to form a biofilm (perhaps influenced by specific oligotypes), creates a lower redox potential in the vaginal microbiome. This alteration would then cause a marked decrease in lactobacilli and an increase in other BVAB that are normally present in very low concentrations, leading to the BV syndrome. Determining the exact etiology of the agent(s) causing a shift from optimal to abnormal vaginal flora and BV is vital for appropriate treatment and prevention of adverse outcomes. With increasing use of molecular methods, identification of vaginal microorganisms (some uncultivable) to the species level in women with BV has become more feasible. This study will seek to further investigate BV pathogenesis. We hypothesize that sexual exposure to Gardnerella vaginalis is the inciting event leading to the complex changes in vaginal flora associated with BV. If Gardnerella vaginalis is the initial insult, then its appearance and establishment in the vaginal microbiome will be seen in women who develop incident BV prior to increases in other BV-associated bacteria.

Only African American women will be enrolled in this protocol as differences in the composition of vaginal microbial communities of women with and without BV of different racial and ethnic groups have been noted which could confound the results of this study.

ELIGIBILITY:
Screening Inclusion Criteria:

1. African American race
2. Female Gender
3. Age 18-45 years
4. History of sexual activity (oral, vaginal, and/or anal) with a female sexual partner during the past 12 months
5. Current female sexual partner
6. English speaking
7. Ability to give written informed consent

Screening Exclusion Criteria:

1. Use of antimicrobials (oral and/or vaginal) within the past 14 days
2. Known HIV
3. Known pregnancy
4. Currently on menstrual period

Enrollment Inclusion Criteria:

1. No Amsel criteria (i.e. patient currently asymptomatic from vaginal discharge standpoint, has normal vaginal pH, negative whiff test, and no clue cells on saline microscopy)
2. Nugent score of 0-3 with no Gardnerella vaginalis morphotypes noted on Gram stain

Enrollment Exclusion Criteria:

1. Presence of current vaginal infections (i.e. trichomoniasis or symptomatic vaginal yeast infection)
2. Pregnancy

   * Reasons for Subsequent Participant Discontinuation after Initial Enrollment**:

(1) Duplicate Nugent score reading > 3 (2) Concurrent trichomonas diagnosis - as determined by nucleic acid amplification testing results

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Sexually active African American women who have sex with women with normal vaginal flora at baseline (determined based on 0/4 Amsel criteria and a normal Nugent score of 0-3 with no Gardnerella vaginalis morphotypes noted on vaginal Gram stain) will be followed prospectively over a 90 day time period for the development of incident BV.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2014-09; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Development of incident BV | 90 days
  Based on 3 consecutive days of Nugent score readings of 7-10 (vaginal Gram stain result)

SECONDARY OUTCOMES:
Development of vaginal symptoms | 90 days
  vaginal discharge, odor, itch based on participant daily diary information (study questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Christina A Muzny, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with statisticians at the University of Mississippi Medical center for statistical analysis.

REFERENCES:
- [Background] Schwebke JR, Muzny CA, Josey WE. Role of Gardnerella vaginalis in the pathogenesis of bacterial vaginosis: a conceptual model. J Infect Dis. 2014 Aug 1;210(3):338-43. doi: 10.1093/infdis/jiu089. Epub 2014 Feb 7. PMID 24511102
- [Background] Muzny CA, Schwebke JR. Gardnerella vaginalis: Still a Prime Suspect in the Pathogenesis of Bacterial Vaginosis. Curr Infect Dis Rep. 2013 Apr;15(2):130-5. doi: 10.1007/s11908-013-0318-4. PMID 23371405
- [Background] Muzny CA, Sunesara IR, Kumar R, Mena LA, Griswold ME, Martin DH, Lefkowitz EJ, Schwebke JR, Swiatlo E. Characterization of the vaginal microbiota among sexual risk behavior groups of women with bacterial vaginosis. PLoS One. 2013 Nov 13;8(11):e80254. doi: 10.1371/journal.pone.0080254. eCollection 2013. PMID 24236175
- [Background] Muzny CA, Sunesara IR, Griswold ME, Kumar R, Lefkowitz EJ, Mena LA, Schwebke JR, Martin DH, Swiatlo E. Association between BVAB1 and high Nugent scores among women with bacterial vaginosis. Diagn Microbiol Infect Dis. 2014 Dec;80(4):321-3. doi: 10.1016/j.diagmicrobio.2014.09.008. Epub 2014 Sep 16. PMID 25262105
- [Background] Schwebke JR, Muzny CA, Josey WE. Reply to Hickey and Forney. J Infect Dis. 2014 Nov 15;210(10):1683-4. doi: 10.1093/infdis/jiu304. Epub 2014 May 22. No abstract available. PMID 24855685
- [Background] Muzny CA, Sunesara IR, Austin EL, Mena LA, Schwebke JR. Bacterial vaginosis among African American women who have sex with women. Sex Transm Dis. 2013 Sep;40(9):751-5. doi: 10.1097/OLQ.0000000000000004. PMID 23949590
- [Background] Muzny CA, Schwebke JR. Editorial commentary: women who have sex with women: a unique population for studying the pathogenesis of bacterial vaginosis. Clin Infect Dis. 2015 Apr 1;60(7):1054-6. doi: 10.1093/cid/ciu1132. Epub 2014 Dec 16. No abstract available. PMID 25516182
- [Background] Muzny CA, Schwebke JR. Biofilms: An Underappreciated Mechanism of Treatment Failure and Recurrence in Vaginal Infections. Clin Infect Dis. 2015 Aug 15;61(4):601-6. doi: 10.1093/cid/civ353. Epub 2015 May 1. PMID 25935553
- [Background] Muzny CA, Schwebke JR. Accuracy of Self-Report of Sexual Activity among Adolescent Girls: Implications for Interpretation of Vaginal Flora Patterns. mBio. 2015 Jun 23;6(3):e00819. doi: 10.1128/mBio.00819-15. No abstract available. PMID 26106081
- [Background] Muzny CA, Blanchard E, Taylor CM, Aaron KJ, Talluri R, Griswold ME, Redden DT, Luo M, Welsh DA, Van Der Pol WJ, Lefkowitz EJ, Martin DH, Schwebke JR. Identification of Key Bacteria Involved in the Induction of Incident Bacterial Vaginosis: A Prospective Study. J Infect Dis. 2018 Aug 14;218(6):966-978. doi: 10.1093/infdis/jiy243. PMID 29718358
- [Background] Van Der Pol WJ, Kumar R, Morrow CD, Blanchard EE, Taylor CM, Martin DH, Lefkowitz EJ, Muzny CA. In Silico and Experimental Evaluation of Primer Sets for Species-Level Resolution of the Vaginal Microbiota Using 16S Ribosomal RNA Gene Sequencing. J Infect Dis. 2019 Jan 7;219(2):305-314. doi: 10.1093/infdis/jiy508. PMID 30535155
- [Background] Olson KM, Boohaker LJ, Schwebke JR, Aslibekyan S, Muzny CA. Comparisons of vaginal flora patterns among sexual behaviour groups of women: implications for the pathogenesis of bacterial vaginosis. Sex Health. 2018 Feb;15(1):61-67. doi: 10.1071/SH17087. PMID 29212588